CLINICAL TRIAL: NCT07376161
Title: The Effect of Pulmonary Rehabilitation on Inflammation and Oxidative Stress in COPD
Brief Title: Inflammation and Oxidative Stress in COPD
Status: Enrolling by invitation | Type: Observational
Sponsor: Deniz Bilici (Other)
Responsible Party: Sponsor-Investigator, Deniz Bilici, MD, Istanbul Medeniyet University
Organization: Istanbul Medeniyet University (Other)
Other Study IDs: 23.10.2025; 2025/0255
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Inflamation; COPD; Oxidative Stress; Pulmonary Rehabilitation
Keywords: COPD; Oxidative Stress; Inflamation; Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Biospecimen Retention: Samples Without DNA — Peripheral venous blood samples will be collected before and after the pulmonary rehabilitation program. Serum samples will be separated and stored for the analysis of inflammatory and oxidative stress biomarkers, including IL-6, TNF-α, IL-33, and NRF-2-related parameters. No DNA extraction or genetic testing will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation — Participants will undergo a standardized, supervised pulmonary rehabilitation program consisting of exercise training, breathing exercises, and patient education. The program will include aerobic exercise training (treadmill or cycle ergometer), strength training of upper and lower limb muscles, and respiratory muscle training, conducted under the supervision of a multidisciplinary rehabilitation team. Sessions will be performed multiple times per week over a predefined program duration. The intervention will be applied in addition to standard pharmacological treatment, with no changes to maintenance medications during the study period.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a leading cause of morbidity and mortality worldwide, characterized by persistent airflow limitation, chronic inflammation, and increased oxidative stress. Despite optimal pharmacological treatment, many patients continue to experience symptoms, reduced exercise capacity, and frequent exacerbations. Pulmonary rehabilitation (PR) is an evidence-based, non-pharmacological intervention that improves symptoms, functional capacity, quality of life, and survival in patients with COPD; however, its biological effects on inflammatory and oxidative stress pathways remain insufficiently defined.

This study aims to evaluate the effects of pulmonary rehabilitation on systemic inflammation and oxidative stress in patients with stable COPD. Serum levels of pro-inflammatory cytokines (IL-6, TNF-α) and the epithelial alarmin IL-33, which is released in response to airway epithelial injury, as well as NRF-2 gene and/or protein expression as a key regulator of antioxidant defense, will be measured before and after a standardized pulmonary rehabilitation program. By assessing changes in these biomarkers, this study seeks to determine whether pulmonary rehabilitation exerts disease-modifying effects beyond symptomatic improvement and functional outcomes.

The findings are expected to provide novel insights into the biological mechanisms of pulmonary rehabilitation and to support its role as a targeted, cost-effective intervention in the comprehensive management of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-80 years with a diagnosis of stable chronic obstructive pulmonary disease (COPD)
* Airflow limitation defined according to GOLD criteria (FEV₁/FVC < 70% and FEV₁ < 70% predicted)
* Former smokers with a smoking history of at least 10 pack-years
* Clinically stable disease at the time of enrollment
* Ability and willingness to participate in the pulmonary rehabilitation program
* Provision of written informed consent

Exclusion Criteria:

* Current smokers
* History of acute COPD exacerbation or respiratory infection within the past 6 weeks
* Presence of other chronic lung diseases (e.g., bronchiectasis, interstitial lung disease, asthma)
* Active malignancy
* Severe or uncontrolled cardiovascular disease, including recent acute myocardial infarction or malignant arrhythmias
* Neurological, orthopedic, or psychiatric conditions that preclude objective functional assessment or participation in exercise training
* Use of antioxidant or vitamin supplementation within the past 4 weeks
* Determination by a cardiologist that participation in an exercise-based rehabilitation program is not medically appropriate

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 40 to 80 years with a diagnosis of stable chronic obstructive pulmonary disease (COPD), defined according to the GOLD criteria (FEV₁/FVC < 70% and FEV₁ < 70% predicted), who are former smokers with a smoking history of at least 10 pack-years, and who are referred to the pulmonary rehabilitation program of our institution, will be consecutively enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Inflammatory and Oxidative Stress Biomarkers After Pulmonary Rehabilitation in COPD Patients | Baseline (before pulmonary rehabilitation) and after 8 weeks of pulmonary rehabilitation
  Primary outcome is the change in serum levels of inflammatory and oxidative stress biomarkers following the pulmonary rehabilitation program in patients with stable COPD. Serum concentrations of IL-6, TNF-α, and IL-33, as well as NRF-2 gene and/or protein expression, will be measured before and after the intervention to evaluate the biological effects of pulmonary rehabilitation on systemic inflammation and oxidative stress.

SECONDARY OUTCOMES:
Association Between Changes in Inflammatory and Oxidative Stress Biomarkers and Clinical and Functional Outcomes After Pulmonary Rehabilitation | Baseline (before pulmonary rehabilitation) and after 8 weeks of pulmonary rehabilitation
  Secondary outcome is the relationship between levels and changes in inflammatory and oxidative stress biomarkers and changes in clinical and functional parameters following pulmonary rehabilitation in patients with stable COPD. Changes in serum IL-6, TNF-α, IL-33, and NRF-2-related parameters will be correlated with post-rehabilitation changes in dyspnea severity, exercise capacity, and health-related quality of life measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
All IPD used in the results publication

REFERENCES:
- [Result] Joppa P, Petrasova D, Stancak B, Dorkova Z, Tkacova R. Oxidative stress in patients with COPD and pulmonary hypertension. Wien Klin Wochenschr. 2007;119(13-14):428-34. doi: 10.1007/s00508-007-0819-y. PMID 17671825
- [Result] Celli BR, Anzueto A, Singh D, Hanania NA, Fabbri L, Martinez FJ, Soler X, Djandji M, Jacob-Nara JA, Rowe PJ, Deniz Y, Radwan A. The Emerging Role of Alarmin-Targeting Biologics in the Treatment of Patients With COPD. Chest. 2025 May;167(5):1346-1355. doi: 10.1016/j.chest.2024.09.049. Epub 2024 Dec 2. PMID 39631681
- [Result] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Result] Mosher CL, Nanna MG, Jawitz OK, Raman V, Farrow NE, Aleem S, Casaburi R, MacIntyre NR, Palmer SM, Myers ER. Cost-effectiveness of Pulmonary Rehabilitation Among US Adults With Chronic Obstructive Pulmonary Disease. JAMA Netw Open. 2022 Jun 1;5(6):e2218189. doi: 10.1001/jamanetworkopen.2022.18189. PMID 35731514
- [Result] Pehlivan E, Yazar E, Balci A, Kilic L. Comparison of Compliance Rates and Treatment Efficiency in Home-Based with Hospital-Based Pulmonary Rehabilitation in COPD. Turk Thorac J. 2019 Jul 1;20(3):192-197. doi: 10.5152/TurkThoracJ.2019.18060. Print 2019 Jul. PMID 31479415
- [Result] Pehlivan E, Yazar E, Balci A, Turan D, Demirkol B, Cetinkaya E. A comparative study of the effectiveness of hospital-based versus home-based pulmonary rehabilitation in candidates for bronchoscopic lung volume reduction. Heart Lung. 2020 Nov-Dec;49(6):959-964. doi: 10.1016/j.hrtlng.2020.06.011. Epub 2020 Jul 21. PMID 32709500
- [Result] Ozmen I, Yildirim E, Ozturk M, Ocakli B, Yildiz R, Aydin R, Karakis M, Yilmaz O, Aksoy E. Pulmonary Rehabilitation Reduces Emergency Admission and Hospitalization Rates of Patients with Chronic Respiratory Diseases. Turk Thorac J. 2018 Sep 13;19(4):170-175. doi: 10.5152/TurkThoracJ.2018.17089. Print 2018 Oct. PMID 30322439
- [Result] Pinho RA, Chiesa D, Mezzomo KM, Andrades ME, Bonatto F, Gelain D, Dal Pizzol F, Knorst MM, Moreira JC. Oxidative stress in chronic obstructive pulmonary disease patients submitted to a rehabilitation program. Respir Med. 2007 Aug;101(8):1830-5. doi: 10.1016/j.rmed.2007.02.004. Epub 2007 Mar 26. PMID 17376663
- [Result] Mercken EM, Hageman GJ, Schols AM, Akkermans MA, Bast A, Wouters EF. Rehabilitation decreases exercise-induced oxidative stress in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 Oct 15;172(8):994-1001. doi: 10.1164/rccm.200411-1580OC. Epub 2005 Jul 22. PMID 16040783
- [Result] Beykumul A, Ersoy Y, Gulbas G, Neselioglu S. Can Blood Biomarkers Be Used to Assess Oxidative Stress in COPD Patients After Pulmonary Rehabilitation. Int J Chron Obstruct Pulmon Dis. 2023 Oct 5;18:2179-2186. doi: 10.2147/COPD.S400415. eCollection 2023. PMID 37818173
- [Result] Zhao X, Zhang Q, Zheng R. The interplay between oxidative stress and autophagy in chronic obstructive pulmonary disease. Front Physiol. 2022 Sep 26;13:1004275. doi: 10.3389/fphys.2022.1004275. eCollection 2022. PMID 36225291
- [Result] Cazzola M, Page CP, Wedzicha JA, Celli BR, Anzueto A, Matera MG. Use of thiols and implications for the use of inhaled corticosteroids in the presence of oxidative stress in COPD. Respir Res. 2023 Jul 31;24(1):194. doi: 10.1186/s12931-023-02500-8. PMID 37517999
- [Result] Miklos Z, Horvath I. The Role of Oxidative Stress and Antioxidants in Cardiovascular Comorbidities in COPD. Antioxidants (Basel). 2023 May 31;12(6):1196. doi: 10.3390/antiox12061196. PMID 37371927
- [Result] Stockley JA, Walton GM, Lord JM, Sapey E. Aberrant neutrophil functions in stable chronic obstructive pulmonary disease: the neutrophil as an immunotherapeutic target. Int Immunopharmacol. 2013 Dec;17(4):1211-7. doi: 10.1016/j.intimp.2013.05.035. Epub 2013 Aug 27. PMID 23994347
- [Result] Zinellu E, Zinellu A, Fois AG, Pau MC, Scano V, Piras B, Carru C, Pirina P. Oxidative Stress Biomarkers in Chronic Obstructive Pulmonary Disease Exacerbations: A Systematic Review. Antioxidants (Basel). 2021 Apr 29;10(5):710. doi: 10.3390/antiox10050710. PMID 33946941
- [Result] Domej W, Oettl K, Renner W. Oxidative stress and free radicals in COPD--implications and relevance for treatment. Int J Chron Obstruct Pulmon Dis. 2014 Oct 17;9:1207-24. doi: 10.2147/COPD.S51226. eCollection 2014. PMID 25378921
- [Result] Barnes PJ. Oxidative Stress in Chronic Obstructive Pulmonary Disease. Antioxidants (Basel). 2022 May 13;11(5):965. doi: 10.3390/antiox11050965. PMID 35624831
- [Result] Katerji M, Filippova M, Duerksen-Hughes P. Approaches and Methods to Measure Oxidative Stress in Clinical Samples: Research Applications in the Cancer Field. Oxid Med Cell Longev. 2019 Mar 12;2019:1279250. doi: 10.1155/2019/1279250. eCollection 2019. PMID 30992736
- [Result] Noguera A, Batle S, Miralles C, Iglesias J, Busquets X, MacNee W, Agusti AG. Enhanced neutrophil response in chronic obstructive pulmonary disease. Thorax. 2001 Jun;56(6):432-7. doi: 10.1136/thorax.56.6.432. PMID 11359957
- [Result] Troosters T, Janssens W, Demeyer H, Rabinovich RA. Pulmonary rehabilitation and physical interventions. Eur Respir Rev. 2023 Jun 7;32(168):220222. doi: 10.1183/16000617.0222-2022. Print 2023 Jun 30. PMID 37286219